## Remote Ischemic Preconditioning and Contrast-Induced Acute Kidney Injury in patients undergoing elective percutaneous coronary intervention

Karolina Stokfisz , MD, Anna Ledakowicz-Polak , MD, PhD,
Michal Kidawa , MD, PhD, Marzenna Zielinska , MD, PhD

ID: RNN/219/13/KE NCT03761368

Corresponding author: Karolina Stokfisz, Intensive Cardiac Therapy Clinic, Department of Invasive Cardiology and Electrocardiology, Medical University of Lodz, Pomorska 251, 2-213 Lodz, Poland, Tel/Fax. +48-42-201 42 60, e-mail: stokfisz.karolina@gmail.com

Running title: Stokfisz et al. RIPC and CI-AKI in patients undergoing elective PCI

## **Statistical Analysis Plan**

We will perform statistical analysis using the STATISTICA 12.5 (StatSoft Inc., Tulsa, OK, USA). For all the tests we will use p = 0.05 as the statistical significance level. Categorical variables will be summarized as frequencies with percentage. Shapiro—Wilk test will be use to assess the normal distribution of variables. Non-parametric statistics will be use when variables had other than normal distribution. Continuous variables with other than normal distribution will be expressed as medians quartile 25 (Q25), quartile 75 (Q75) with interquartile range (IQR). Correlations will be assessed by using Spearman's rank correlation coefficient. Differences between continuous variables will be compared by using Mann—Whitney U test, whereas differences between categorical variables will be compared by chi-squared test with Yates's correction for continuity. The Wilcoxon signed-rank test will be use to compare repeated measurements. To assess the suitability of NGAL values in CI-AKI occurrence probability estimation, the receiver operating characteristic (ROC) curve analysis will be performed.